

### Determination of Postoperative Stroke Incidence in Patients With and Without the Use of Epiaortic Ultrasound in Coronary Artery Bypass Grafting Surgery

Brief Title: Postoperative Stroke and Epiaortic Ultrasound in CABG

Document Date: July 13, 2025



## INFORMED CONSENT FORM FOR CORONARY ARTERY BYPASS GRAFT (CABG)

| Patient's: |
|-----------------------------------------------------------------------|
| File No: |
| Name: |
| Surname: |
| Date of Birth: |
| PROPOSED TREATMENT |
| My doctor |
| Coronary Artery Bypass Graft(s) (CABG) surgery due to the presence of |

This procedure involves bypassing the blocked or narrowed blood vessels in the heart using veins and/or arteries harvested from other parts of the body.

Under general anesthesia, the sternum is cut and the chest is opened. If the surgeon deems appropriate and with prior patient consent, the surgery may be performed through a smaller incision or between the ribs. The blood vessels to be used as grafts (internal thoracic artery, arm artery, saphenous vein from the leg, or another vessel) are prepared.

The surgeon opens the chest and uses a machine (heart-lung machine) to take over the function of the heart and lungs. Once connected, the heart and lungs are taken out of operation. The body is cooled to protect vital tissues and organs. The heart is stopped while the grafts are sutured in place. In some cases, the surgeon may choose to perform the grafts without stopping the heart or using the bypass machine (your surgeon will inform you if this is the case). Occasionally, although the surgery is started without the pump, it may become necessary to use it.

One or more chest tubes may be temporarily placed in the chest cavity to allow the lungs to reexpand and drain any accumulated fluid. One or two pacing wires may be attached to the heart to

monitor and control the heart rhythm postoperatively. The sternum is wired shut, and the skin is closed.



### RISKS

The purpose of this explanation is not to scare or worry you, but to provide you with informed knowledge about your surgery and its risks.

These are commonly seen risks; rarer complications not mentioned here may also occur. Please ask your surgeon if you have any general or specific questions.

These risks may occur with any anesthetic. You may experience side effects from any of the medications used. Common ones include dizziness, nausea, skin rashes, and constipation.

The planned surgery (Coronary artery bypass graft surgery) has the following risks and limitations:

- There is a small risk of death.
- Bleeding at the surgical site may occur; if uncontrolled, reoperation may be required.
- Parts of the lungs may collapse, increasing the risk of lung infections, possibly requiring
  physiotherapy and antibiotics. Time on the ventilator may be prolonged, and ICU stay
  extended.
- Temporary or permanent brain function impairment may occur during surgery. Vegetative state may develop postoperatively.
- If your heart does not function adequately after the operation, a support device may be inserted through the groin vessels. This may cause circulatory problems in the leg, requiring surgical intervention.
- Rarely, kidney failure may develop, requiring temporary or permanent dialysis.
- Wounds may become infected, showing redness, pain, and swelling, possibly requiring antibiotics. In some cases, the wound may need to be reopened and reoperated.
- The sternum may fail to heal due to infection or improper movement, necessitating reoperation.
- Palpitations, especially rapid rhythm called atrial fibrillation, may occur. This can be managed with medication or electrical intervention if needed.
- Deep vein thrombosis (DVT) may develop in the legs, with pain and swelling. A clot may dislodge and travel to the lungs (pulmonary embolism), potentially causing shortness of breath and, rarely, death.
- Stomach bleeding may occur as a side effect of surgical stress or medication.
- Embolic particles from the main artery leaving the heart may cause intestinal infarctions, which may require emergency surgery due to this life-threatening complication.
- Temporary postoperative confusion may occur for a few days.



- Blood transfusion may be necessary.
- Fluid accumulation around the lungs or heart may require needle drainage.
- Bleeding or fluid collection may develop at the surgical site. While this may be reabsorbed naturally, reoperation is rarely needed.

These risks are increased if you smoke, have chronic lung disease, obesity, diabetes, high blood pressure, or known heart disease.

# INDIVIDUAL RISKS After deciding to undergo this surgery, the following risks and complications may arise based on your personal characteristics:

| <br>• • • • |
|-------------|

### PATIENT DECLARATION

- My surgeon has informed me about the procedure and alternative treatment options and answered my questions on specific concerns.
- After deciding on surgery, my surgeon informed me about risks and complications that may arise based on my personal characteristics.
- I accept that additional procedures deemed necessary by my surgeon during surgery may be performed.
- I consent to blood transfusion if required.
- I agree that any tissue removed during the procedure may be disposed of by hospital authorities. I understand that some samples may be retained as part of my hospital record.
- I accept that the planned surgical procedure will be carried out by the doctor ...... and their team.
- I understand that photographs and videos may be taken for medical education purposes
  during the procedure, that they will be used solely for educational purposes by medical
  personnel, and that my identity will not be revealed.
- I have received a copy of this form for my records.
- If a needle or sharp object injures a team member during surgery, I agree to provide an additional blood sample for screening of HIV and other bloodborne diseases for research purposes. I understand that I will be informed and advised as soon as possible after surgery if this occurs.
- I have read and understood all 3 (three) pages of this consent form.



PATIENT NAME

**DATE** 

PATIENT SIGNATURE

REPRESENTATIVE'S DECLARATION (If the patient is not able to provide consent)

I have read and understood the explanations regarding the procedure, its consequences, and risks. As the patient is not in a condition to provide consent, I authorize the surgery on their behalf.

REPRESENTATIVE'S NAME

**DATE** 

**SIGNATURE** 

### PHYSICIAN'S DECLARATION

I declare that I have provided the necessary explanation regarding the procedure and its consequences, and I have informed the patient about the possible risks. I gave the patient the opportunity to ask questions and answered them.

DOCTOR'S NAME

DATE

DOCTOR'S SIGNATURE

### WITNESS DECLARATION (Preferably a relative)

I confirm that I witnessed the explanation of this form and the conversation between the doctor and the patient.

WITNESS NAME

**DATE** 

WITNESS SIGNATURE